CLINICAL TRIAL: NCT04316091
Title: A Phase I Clinical Trial of Neoadjuvant Chemotherapy With/Without Superparamagnetic Iron Oxide Nanoparticles and Spinning Magnetic Field for Patients With Osteosarcoma
Brief Title: A Phase I Clinical Trial of Neoadjuvant Chemotherapy With/Without SPIONs/SMF for Patients With Osteosarcoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YANWQ004
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): neoadjuvant chemotherapy+SPIONs/SMF
  Interventions: Drug: neoadjuvant chemotherapy+SPIONs/SMF
- Control group (Sham Comparator): neoadjuvant chemotherapy
  Interventions: Drug: neoadjuvant chemotherapy

INTERVENTIONS:
Drug: neoadjuvant chemotherapy+SPIONs/SMF — Intratumoral injection of SPIONs, followed by SMF, combined with conventional neoadjuvant chemotherapy
  Arms: Experimental group
Drug: neoadjuvant chemotherapy — Conventional neoadjuvant chemotherapy only
  Arms: Control group

SUMMARY:
Osteosarcoma is the most common primary malignant bone tumor that mainly occurs in children and adolescents. Combined surgical resection and intensive chemotherapy has improved the 5-year overall survival rate (from 51 to 75%). However, drug-induced side effects and tumor recurrence after surgery reduce patient quality of life and cut down the patient survival rate. Superparamagnetic Iron Oxide Nanoparticles (SPIONs)/Spinning Magnetic Field (SMF) and neoadjuvant chemotherapy may increase the cancer cell killing and complete tumor shrinkage preserving local structures and functions of patients who cannot receive limb retention treatment.

DETAILED DESCRIPTION:
This study aims to evaluate the safety, efficacy, and tolerability of SPIONs/SMF in combination with neoadjuvant chemotherapy in osteosarcoma patients. They will receive intratumoral injection of SPIONs every other day for 3 times, followed by SMF for 2 hours every two days, and up to completion of 30 days, and conventional neoadjuvant chemotherapy from day 1. The sponsor hypothesizes that SPIONs/SMF will act synergistically with neoadjuvant chemotherapy to increase the cancer cell killing, to increase the local efficacy of neoadjuvant chemotherapy, and to improve the ratio of limb retention. Then, all patients will be followed every 8 weeks, for the safety evaluation and cancer disease status until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Biopsy-confirmed cancer diagnosis
* Has at least one tumor lesion that can be accurately measured according to RECIST 1.1. and is amenable for intratumoral injection
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy >12 weeks
* Karnofsky performance status (KPS) ≥ 70
* Adequate function of organs and bone marrow
* Negative pregnancy test ≤ 7 days prior to SPIONs injection

Exclusion Criteria:

* Symptomatic central nervous system metastases and/or carcinomatous meningitis
* Known HIV or active hepatitis B/C infection
* Active infection requiring systemic treatment
* Received a live virus vaccine within 30 days prior to study treatment
* History of pneumonitis that required steroids or with current pneumonitis
* Has received prior systemic anti-neoplastic therapy, within 4 weeks prior to SPIONs injection
* Clinically significant cardiac arrhythmias
* Class III or IV Congestive Heart Failure as defined by the New York Heart Association functional classification system < 6 months prior to screening
* A pregnant or nursing female, or women of child-bearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Any condition for which participation would not be in the best interest of the participant
* Patients unable to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures or those with severe psychiatric illness/social situations that would limit compliance with study requirements
* Patients participating in another clinical investigation at the time of signature of the informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Determination of the Recommended Dose | 36 Months
  Determination of dose-limiting toxicities (DLTs), the maximum tolerated dose (MTD) (if possible), and recommended Phase 2 doses (RP2Ds)

SECONDARY OUTCOMES:
Evaluation of the anti-tumor response of neoadjuvant chemotherapy±SPIONs/SMF | 36 Months
  Evaluation of the Objective Response Rate: complete or partial response, as defined by RECIST 1.1
Assessment of the safety and feasibility of neoadjuvant chemotherapy±SPIONs/SMF | 36 Months
  Assessment of the number of participants with related late onset toxicities defined as any Grade ≥3 adverse event (AE) occurring after the end of treatment (EOT) visit
Evaluation of the body kinetic profile of intratumorally injected neoadjuvant chemotherapy±SPIONs/SMF | 36 Months
  Evaluation of the time-course dependent accumulation (μg/dL) of iron in blood and urine following SPIONs intratumoral injection